CLINICAL TRIAL: NCT06061354
Title: Bone Microarchitecture and Implant Stabilization in Atrophic Jaws Reconstructed With Bone Grafts Treated With Teriparatide
Brief Title: Teriparatide on Maxillary Sinus Floor Osseointegration
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Valparaiso (Other)
Collaborators: Universidade Federal Fluminense (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEC 256-22
Record Dates: First submitted 2023-09-08; First posted 2023-09-29 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Bone Regeneration
Keywords: teriparatide; Bio-Oss®; bone graft; dental implants; maxillary sinus augmentation; bone regeneration
MeSH Terms: interventions — Teriparatide; Sinus Floor Augmentation; Bone Transplantation; Bio-Oss

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Teriparatide (Experimental): Access to the maxillary sinus will be done through osteotomy, using a piezosurgery . Subsequently, the Schneider's membrane will be carefully lifted and, according to the randomization process, the graft material Bio-Oss® mixed with Forteo® will be delivered for placement on the sinus floor maxilla below Schneider's membrane.
  Next, the access window to the maxillary sinus and Schneider's membrane will be protected. The mucoperiosteal flap will be repositioned and closed
  Interventions: Drug: Teriparatide; Procedure: Maxillary Sinus Augmentation; Procedure: Dental Implant Installation; Combination Product: Bone graft
- Placebo (Placebo Comparator): Access to the maxillary sinus will be done through osteotomy, using a piezosurgery . Subsequently, the Schneider's membrane will be carefully lifted and, according to the randomization process, the graft material, Bio-Oss® mixed with saline solution, will be delivered for placement on the sinus floor maxilla below Schneider's membrane.
  Next, the access window to the maxillary sinus and Schneider's membrane will be protected. The mucoperiosteal flap will be repositioned and closed
  Interventions: Procedure: Maxillary Sinus Augmentation; Procedure: Dental Implant Installation; Combination Product: Bone graft

INTERVENTIONS:
Drug: Teriparatide — mixture of 20μg of teriparatide, 0.64ml of saline solution with 1g of Bio -Oss® or 1g of Bio-Oss® will be mixed with 0.72ml of saline solution.
  Other Names: Teriparatide Pen Injector [Forteo]
  Arms: Teriparatide
Procedure: Maxillary Sinus Augmentation — Local anesthesia will be performed, mucoperiosteal flap will be raised to access the anterior wall of the maxillary sinus. Access to the maxillary sinus will be done through osteotomy, using a piezosurgery under irrigation with saline solution. Subsequently, the Schneider's membrane will be carefully lifted and, according to the randomization process, the graft material (Bio-Oss® mixed with saline solution or Bio-Oss® mixed with Forteo®) will be delivered for placement on the sinus floor maxilla below Schneider's membrane.Next, the access window to the maxillary sinus and Schneider's membrane will be protected. The mucoperiosteal flap will be repositioned and closed.
Procedure: Dental Implant Installation — Local anesthesia will be performed a mucoperiosteal flap will be raised in the area for implant placement and a bone core 10 mm high and 2 mm in diameter will be removed with a 2 mm trephine bur. The bone biopsied through this nucleus is part of the region where the implant will be installed, and the height of the sample depends on the surgical planning carried out previously (3-month radiographic control). The sequence of drills to place the implant will continue, installation of the implant itself and, finally, verification of the insertion torque and measurement of the resonance frequency in the already installed implant. The mucoperiosteal flap must be repositioned and sutured.
Combination Product: Bone graft — One arm:mixture of 20μg of teriparatide, 0.64ml of saline solution with 1g of Bio -Oss® In other arm: 1g of Bio-Oss® will be mixed with 0.72ml of saline solution.
  Other Names: Bio-Oss®

SUMMARY:
The aim of this triple blind randomized controlled trial will be to analyze the effect of a dose of teriparatide combined with a xenograft on bone augmentation of the maxillary sinus, to observe the microarchitecture of the newly formed bone and the primary and late stability of implants placed on these grafts. The sample is composed of 42 participants who have a clinical indication for maxillary sinus floor augmentation with bone grafting due to residual bone height less than or equal to 5mm for the installation of dental implants. Each side will be grafted with Bio-Oss® or Bio-Oss® combined with 1 dose (20 µg) of teriparatide (Forteo®). Three months after grafting, at the time of placement of dental implants, bone biopsies will be obtained using a short 2mm trephine bur. These bone cores will be submitted to histological and histomorphometric analysis. The stability of the implants will be measured, at the time of their installation, through the insertion torque, and through the use of resonance frequency equipment (Ostell®) in three moments: immediately and at 3 and 6 months after the installation of the dental implants.

ELIGIBILITY:
Inclusion Criteria:

* Pneumatization of a maxillary sinus with a residual ridge ≤ 5 mm in height (according to baseline conebeam tomograph).
* Must sign an informed consent to participate in this study.

Exclusion Criteria:

* Residual ridges less than 4 mm in height.
* Uncontrolled systemic disease (ASA 3, 4, 5, and 6)
* Presenting with osteoporosis or any disease of bone metabolism.
* Having received radiotherapy.
* Cancer.
* Any systemic condition that affects calcium absorption.
* Kidney disease.
* Coagulation disorders.
* History of sinusitis.
* Maxillary sinus pathology.
* Heavy smoking (> 1 pack per day).
* Drug or alcohol users.
* Pregnancy.
* Treatment with drugs that affect bone metabolism.
* Treatment with immunosuppressants.
* Allergies.
* Uncontrolled periodontal pathology.
* Tooth extractions in the last three months.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-08-23 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Histology | 3 months
  osteoblasts/mm2

SECONDARY OUTCOMES:
Histomorphometry | 3 months
  Describe de presence of following parameters: necrosis, inflammation, vascularization and angiogenesis, fibrosis, presence of medullary adipose tissue, new bone formation and foreign body reaction

OTHER OUTCOMES:
implant stability coefficient (ISQ) | 6 months
  The implant stability coefficient (ISQ) will be evaluated by measuring the resonance frequency and the insertion torque at the time of implant installation. The implanted stability value, evaluated will be measured in two mutually perpendicular directions (distal mesio and palatine bucal). The scale goes from 1 to 100, where higher values indicate greater stability. The acceptable stability range is between 55 and 85 ISQ
Bone Level | 6 months
  Be evaluated using cone beam tomography images, using linear measurement in milimeter (mm) of the floor of the maxillary sinus and should include from the lowest point of the alveolar process to the most superior radiopaque point of the floor of the maxillary sinus exactly in the region where the grafts will be performed and later the installation of the implants.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Seabra Louro, DDS,MSc,PhD, Study Director — Universidade Federal Fluminense
Locations (1):
- Facultad de Odontología, Universidad de Valparaiso, Valparaíso, Región de Valparaíso, Chile

REFERENCES:
- [Background] Miller SC, Hunziker J, Mecham M, Wronski TJ. Intermittent parathyroid hormone administration stimulates bone formation in the mandibles of aged ovariectomized rats. J Dent Res. 1997 Aug;76(8):1471-6. doi: 10.1177/00220345970760080901. PMID 9240383
- [Background] Boabaid F, Berry JE, Koh AJ, Somerman MJ, McCcauley LK. The role of parathyroid hormone-related protein in the regulation of osteoclastogenesis by cementoblasts. J Periodontol. 2004 Sep;75(9):1247-54. doi: 10.1902/jop.2004.75.9.1247. PMID 15515341
- [Background] Jung RE, Cochran DL, Domken O, Seibl R, Jones AA, Buser D, Hammerle CH. The effect of matrix bound parathyroid hormone on bone regeneration. Clin Oral Implants Res. 2007 Jun;18(3):319-25. doi: 10.1111/j.1600-0501.2007.01342.x. Epub 2007 Mar 26. PMID 17386063
- [Background] Liu J, Cao Z, Li C. Intermittent PTH administration: a novel therapy method for periodontitis-associated alveolar bone loss. Med Hypotheses. 2009 Mar;72(3):294-6. doi: 10.1016/j.mehy.2008.10.015. Epub 2008 Nov 30. PMID 19046622
- [Background] Rowshan HH, Parham MA, Baur DA, McEntee RD, Cauley E, Carriere DT, Wood JC, Demsar WJ, Pizarro JM. Effect of intermittent systemic administration of recombinant parathyroid hormone (1-34) on mandibular fracture healing in rats. J Oral Maxillofac Surg. 2010 Feb;68(2):260-7. doi: 10.1016/j.joms.2009.09.045. PMID 20116693
- [Background] Valderrama P, Jung RE, Thoma DS, Jones AA, Cochran DL. Evaluation of parathyroid hormone bound to a synthetic matrix for guided bone regeneration around dental implants: a histomorphometric study in dogs. J Periodontol. 2010 May;81(5):737-47. doi: 10.1902/jop.2010.090562. PMID 20429653
- [Background] Zeng X, He H, Zhang L, Wu Y, Wang Y, Gong P. A potential therapeutic approach to overload-induced bone loss around implant: parathyroid hormone (PTH). Med Hypotheses. 2011 Nov;77(5):701-4. doi: 10.1016/j.mehy.2011.06.016. Epub 2011 Sep 9. PMID 21908105
- [Background] Kuchler U, Luvizuto ER, Tangl S, Watzek G, Gruber R. Short-term teriparatide delivery and osseointegration: a clinical feasibility study. J Dent Res. 2011 Aug;90(8):1001-6. doi: 10.1177/0022034511407920. Epub 2011 May 9. PMID 21555773
- [Background] Ali MN, Kobayashi T, Tanaka M, Ohshima H, Ejiri S, Saito C. Effects of intermittent parathyroid hormone treatment on new bone formation during distraction osteogenesis in the rat mandible. Oral Surg Oral Med Oral Pathol Oral Radiol. 2012 Jul;114(1):e36-42. doi: 10.1016/j.oooo.2011.08.009. Epub 2012 Feb 25. PMID 22727105
- [Background] Aggarwal P, Zavras A. Parathyroid hormone and its effects on dental tissues. Oral Dis. 2012 Jan;18(1):48-54. doi: 10.1111/j.1601-0825.2011.01850.x. Epub 2011 Sep 6. PMID 21895887
- [Background] Wolf M, Lossdorfer S, Abuduwali N, Meyer R, Kebir S, Gotz W, Jager A. Effect of intermittent PTH(1-34) on human periodontal ligament cells transplanted into immunocompromised mice. Tissue Eng Part A. 2012 Sep;18(17-18):1849-56. doi: 10.1089/ten.TEA.2011.0626. Epub 2012 May 21. PMID 22497226
- [Background] Chan HL, McCauley LK. Parathyroid hormone applications in the craniofacial skeleton. J Dent Res. 2013 Jan;92(1):18-25. doi: 10.1177/0022034512464779. Epub 2012 Oct 15. PMID 23071071
- [Background] Kuroshima S, Kovacic BL, Kozloff KM, McCauley LK, Yamashita J. Intra-oral PTH administration promotes tooth extraction socket healing. J Dent Res. 2013 Jun;92(6):553-9. doi: 10.1177/0022034513487558. Epub 2013 Apr 23. PMID 23611925
- [Background] Kuroshima S, Al-Salihi Z, Yamashita J. Parathyroid hormone related to bone regeneration in grafted and nongrafted tooth extraction sockets in rats. Implant Dent. 2013 Feb;22(1):71-6. doi: 10.1097/ID.0b013e318278f94d. PMID 23296032
- [Background] Lima LL, Cesar Neto JB, Cayana EG, Nociti FH Jr, Sallum EA, Casati MZ. Parathyroid hormone (1-34) compensates the negative effect of smoking around implants. Clin Oral Implants Res. 2013 Sep;24(9):1055-9. doi: 10.1111/j.1600-0501.2012.02502.x. Epub 2012 Jun 19. PMID 22712894
- [Background] Tang ZL, Zhang WJ, Wang DX, Chen JM, Ma H, Wu DR. An experimental study addressing the promotion of mandibular defect repair through the intermittent subcutaneous injection of parathyroid hormone. J Oral Maxillofac Surg. 2014 Feb;72(2):419-30. doi: 10.1016/j.joms.2013.07.037. Epub 2013 Sep 24. PMID 24071373
- [Background] Vasconcelos DF, Marques MR, Benatti BB, Barros SP, Nociti FH Jr, Novaes PD. Intermittent parathyroid hormone administration improves periodontal healing in rats. J Periodontol. 2014 May;85(5):721-8. doi: 10.1902/jop.2013.130155. Epub 2013 Jul 29. PMID 23895251
- [Background] Ersan N, van Ruijven LJ, Bronckers AL, Olgac V, Ilguy D, Everts V. Teriparatide and the treatment of bisphosphonate-related osteonecrosis of the jaw: a rat model. Dentomaxillofac Radiol. 2014;43(1):20130144. doi: 10.1259/dmfr.20130144. Epub 2013 Oct 29. PMID 24170800
- [Background] Kakehashi H, Ando T, Minamizato T, Nakatani Y, Kawasaki T, Ikeda H, Kuroshima S, Kawakami A, Asahina I. Administration of teriparatide improves the symptoms of advanced bisphosphonate-related osteonecrosis of the jaw: preliminary findings. Int J Oral Maxillofac Surg. 2015 Dec;44(12):1558-64. doi: 10.1016/j.ijom.2015.07.018. Epub 2015 Aug 21. PMID 26304604
- [Background] Tsunori K. Effects of parathyroid hormone dosage and schedule on bone regeneration. J Oral Sci. 2015 Jun;57(2):131-6. doi: 10.2334/josnusd.57.131. PMID 26062862
- [Background] Otawa M, Tanoue R, Kido H, Sawa Y, Yamashita J. Intermittent administration of parathyroid hormone ameliorates periapical lesions in mice. J Endod. 2015 May;41(5):646-51. doi: 10.1016/j.joen.2014.12.008. Epub 2015 Jan 30. PMID 25649296
- [Background] Keskinruzgar A, Bozdag Z, Aras MH, Demir T, Yolcu U, Cetiner S. Histopathological Effects of Teriparatide in Medication-Related Osteonecrosis of the Jaw: An Animal Study. J Oral Maxillofac Surg. 2016 Jan;74(1):68-78. doi: 10.1016/j.joms.2015.07.005. Epub 2015 Jul 14. PMID 26215490
- [Background] dos Santos RA, Ferreira MS, Mafra CE, Holzhausen M, de Lima LA, Mendes Pannuti C, Cesar Neto JB. Synthetic Parathyroid Hormone May Augment Bone Volume in Autogenous Grafts: A Study in Rats. J Periodontol. 2016 Jan;87(1):66-73. doi: 10.1902/jop.2015.140638. Epub 2015 Sep 25. PMID 26404581
- [Background] Javed F, Al Amri MD, Kellesarian SV, Al-Kheraif AA, Vohra F, Calvo-Guirado JL, Malmstrom H, Romanos GE. Efficacy of parathyroid hormone supplementation on the osseointegration of implants: a systematic review. Clin Oral Investig. 2016 May;20(4):649-58. doi: 10.1007/s00784-015-1691-1. Epub 2015 Dec 22. PMID 26689569
- [Background] Zandi M, Dehghan A, Mohammadi-Mofrad A, Amini P, Vahdatinia F. Short-term perioperative teriparatide therapy for the prevention of medication-related osteonecrosis of the jaw: A randomized, controlled preclinical study in rats. J Craniomaxillofac Surg. 2017 Feb;45(2):275-280. doi: 10.1016/j.jcms.2016.12.010. Epub 2016 Dec 19. PMID 28087282
- [Background] Zandi M, Dehghan A, Zandipoor N, Amini P, Doulati S. Effect of different doses and durations of teriparatide therapy on resolution of medication-related osteonecrosis of the jaw: A randomized, controlled preclinical study in rats. J Craniomaxillofac Surg. 2018 Mar;46(3):466-472. doi: 10.1016/j.jcms.2017.12.027. Epub 2017 Dec 30. PMID 29395991
- [Background] Goker F, Ersanli S, Arisan V, Cevher E, Guzel EE, Issever H, Omer B, Durmus Altun G, Morina D, Ekiz Yilmaz T, Dervisoglu E, Del Fabbro M. Combined effect of parathyroid hormone and strontium ranelate on bone healing in ovariectomized rats. Oral Dis. 2018 Oct;24(7):1255-1269. doi: 10.1111/odi.12895. Epub 2018 Jun 11. PMID 29774969
- [Background] Zandi M, Dehghan A, Amini P, Doulati S, Rezaeian L. Evaluation of the effect of teriparatide therapy on mandibular fracture healing in rats with medication-related osteonecrosis of the jaw. Clin Oral Investig. 2019 Nov;23(11):3987-3993. doi: 10.1007/s00784-019-02830-2. Epub 2019 Feb 4. PMID 30715621
- [Background] Yoshida W, Matsugami D, Murakami T, Bizenjima T, Imamura K, Seshima F, Saito A. Combined effects of systemic parathyroid hormone (1-34) and locally delivered neutral self-assembling peptide hydrogel in the treatment of periodontal defects: An experimental in vivo investigation. J Clin Periodontol. 2019 Oct;46(10):1030-1040. doi: 10.1111/jcpe.13170. PMID 31292977
- [Background] Zandi M, Dehghan A, Gheysari F, Rezaeian L, Mohammad Gholi Mezerji N. Evaluation of teriparatide effect on healing of autografted mandibular defects in rats. J Craniomaxillofac Surg. 2019 Jan;47(1):120-126. doi: 10.1016/j.jcms.2018.11.015. Epub 2018 Nov 23. PMID 30528562
- [Background] de Oliveira D, de Oliveira Puttini I, Silva Gomes-Ferreira PH, Palin LP, Matsumoto MA, Okamoto R. Effect of intermittent teriparatide (PTH 1-34) on the alveolar healing process in orchiectomized rats. Clin Oral Investig. 2019 May;23(5):2313-2322. doi: 10.1007/s00784-018-2672-y. Epub 2018 Oct 6. PMID 30291494
- [Background] Li Y, Chen XY, Tang ZL, Tan JQ, Wang DX, Dong Q. Differences in accelerated tooth movement promoted by recombinant human parathyroid hormone after mandibular ramus osteotomy. Am J Orthod Dentofacial Orthop. 2019 May;155(5):670-680. doi: 10.1016/j.ajodo.2018.06.014. PMID 31053283
- [Background] Zandi M, Dehghan A, Bigonah N, Doulati S, Mohammad Gholi Mezerji N. Histological assessment of the effects of teriparatide therapy on mandibular fracture healing: A preclinical study. J Craniomaxillofac Surg. 2020 Mar;48(3):211-216. doi: 10.1016/j.jcms.2020.01.006. Epub 2020 Jan 21. PMID 32014386
- [Background] Zhang C, Li T, Zhou C, Huang L, Li Y, Wang H, Duan P, Zou S, Mei L. Parathyroid hormone increases alveolar bone homoeostasis during orthodontic tooth movement in rats with periodontitis via crosstalk between STAT3 and beta-catenin. Int J Oral Sci. 2020 Dec 30;12(1):38. doi: 10.1038/s41368-020-00104-2. PMID 33380723
- [Background] Pelled G, Lieber R, Avalos P, Cohn-Schwartz D, Tawackoli W, Roth J, Knapp E, Schwarz EM, Awad HA, Gazit D, Gazit Z. Teriparatide (recombinant parathyroid hormone 1-34) enhances bone allograft integration in a clinically relevant pig model of segmental mandibulectomy. J Tissue Eng Regen Med. 2020 Aug;14(8):1037-1049. doi: 10.1002/term.3075. Epub 2020 Jun 25. PMID 32483878
- [Background] Dam C, Jung UW, Park KM, Huh J, Park W. Effect of teriparatide on early sinus graft healing in the ovariectomized rabbit. Clin Oral Implants Res. 2020 Mar;31(3):264-273. doi: 10.1111/clr.13565. Epub 2020 Jan 3. PMID 31837052
- [Background] Stutz C, Batool F, Petit C, Strub M, Kuchler-Bopp S, Benkirane-Jessel N, Huck O. Influence of parathyroid hormone on periodontal healing in animal models: A systematic review. Arch Oral Biol. 2020 Dec;120:104932. doi: 10.1016/j.archoralbio.2020.104932. Epub 2020 Oct 6. PMID 33113458
- [Background] Emam H, Leach D, Sun Z, Tee BC, Karatas B, Kim DG, Jatana C. The Effect of Parathyroid Hormone Analogues When Added to Mineralized Bone Xenografts. J Oral Implantol. 2020 Aug 1;46(4):372-379. doi: 10.1563/aaid-joi-D-19-00016. PMID 32299092
- [Background] Koca CG, Kosehasanogullari M. Evaluation of single-dose applied teriparatide effect on bone healing with histomorphometric and micro-ct analysis. J Craniomaxillofac Surg. 2021 Feb;49(2):98-103. doi: 10.1016/j.jcms.2020.12.004. Epub 2020 Dec 17. PMID 33384204
- [Background] Jung J, Shim GJ, Kim M, Yoon Y, Kim JE, Jue SS, Al-Nawas B, Kwon YD. Effect and timing of parathyroid hormone analog administration for preventing medication-related osteonecrosis of the jaws in a murine model. J Craniomaxillofac Surg. 2021 Aug;49(8):719-725. doi: 10.1016/j.jcms.2021.02.023. Epub 2021 Feb 26. PMID 33722457
- [Background] Anabtawi M, Tweedale H, Mahmood H. The role, efficacy and outcome measures for teriparatide use in the management of medication-related osteonecrosis of the jaw. Int J Oral Maxillofac Surg. 2021 Apr;50(4):501-510. doi: 10.1016/j.ijom.2020.07.021. Epub 2020 Aug 14. PMID 32800674
- [Background] Ebrahimi S, Navabazam A, Salemi F, Khaleghi F, Barzegar M, Saghafi F, Fallahzadeh H. The efficacy of teriparatide (Cinnopar(R)) on bone repair in mandibular fractures: A single blinded randomized clinical trial. J Craniomaxillofac Surg. 2022 Dec;50(12):923-928. doi: 10.1016/j.jcms.2022.12.002. Epub 2023 Jan 5. PMID 36646571
- [Background] Grossi JRA, Deliberador TM, Giovanini AF, Zielak JC, Sebastiani A, Gonzaga CC, Coelho PG, Zetola AL, Weiss FP, Benalcazar Jalkh EB, Storrer CLM, Witek L. Effects of local single dose administration of parathormone on the early stages of osseointegration: A pre-clinical study. J Biomed Mater Res B Appl Biomater. 2022 Aug;110(8):1806-1813. doi: 10.1002/jbm.b.35038. Epub 2022 Feb 26. PMID 35218605
- [Background] Camili Y, Malkoc S, Taslidere A, Ileri Z, Guler OC. Effects of teriparatide on bone formation in rats with experimentally induced premaxillary expansion. Dental Press J Orthod. 2022 Jul 4;27(3):e2220370. doi: 10.1590/2177-6709.27.3.e2220370.oar. eCollection 2022. PMID 35792789
- [Background] Li Y, Qian Y, Qiao H, Pan W, Xie L, Li Y. Abaloparatide outperforms teriparatide in protecting against alveolar bone loss in experimental periodontitis. J Periodontol. 2023 Feb;94(2):244-255. doi: 10.1002/JPER.22-0211. Epub 2022 Nov 8. PMID 35892139

DOCUMENTS (2):
  • Study Protocol (2023-09-19): https://cdn.clinicaltrials.gov/large-docs/54/NCT06061354/Prot_000.pdf
  • Informed Consent Form (2023-08-28): https://cdn.clinicaltrials.gov/large-docs/54/NCT06061354/ICF_001.pdf